CLINICAL TRIAL: NCT02548819
Title: University Hospital Cardiac Device MR Registry: The Safety of MR Imaging in Patients With Implanted Cardiac Devices
Acronym: CDMR
Status: Completed | Type: Observational
Sponsor: University Health Care System, Augusta, Georgia (Other)
Responsible Party: Principal Investigator, Patrick Aquilina, Physician, Division of Cardiac Electrophysiology, University Health Care System, Augusta, Georgia
Other Study IDs: IORG0000351
Record Dates: First submitted 2015-09-09; First posted 2015-09-14 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: MRI; Pacemaker; Defibrillator

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: MRI — MR imaging of patients with implanted cardiac devices

SUMMARY:
A single-center registry to prospectively evaluate the safety of non-cardiac/non-thoracic magnetic resonance imaging (MRI) in patients with implanted cardiac devices (pacemakers and implantable cardioverter defibrillators).

DETAILED DESCRIPTION:
Evaluation of safety of MR scanning of patients with implanted cardiac devices. Device parameters pre and post MR imaging will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years or older
* Informed consent can be provided by patient or medical power of attorney
* Presence of implanted pacemaker or ICD
* MRI is the diagnostic modality of choice for a specific clinical scenario without acceptable alternative imaging technology as determined by ordering physician
* Non-cardiac/non-thoracic MRI ordered

Exclusion Criteria:

* Presence of metallic objects that represent a contraindication to MR imaging
* Morbid obesity which results in body contact with the magnet façade
* Pacemaker or ICD generator implanted prior to 2002
* ICD patients who are pacing dependent
* Pregnancy
* Device generator at ERI (elective replacement interval)
* Presence of other active implanted medical device
* Presence of abandoned leads (with the exception of post CABG temporary epicardial pacing wires)
* Presence of implanted cardiac device in the abdominal position
* Pacemaker or ICD that is labeled as MRI-Conditional by the FDA
* Pacemaker or ICD implanted less than 6 weeks prior to MRI scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who require MR imaging in the presence of a pacemaker or ICD
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2015-09; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Battery voltage | Immediate
  Change in voltage > 0.04 V
Pacing lead impedance | Immediate
  Change in impedance > 50 Ohms
Shock impedance | Immediate
  Change in impedance > 3 Ohms
P wave amplitude | Immediate
  Decrease in amplitude > 50%
R wave amplitude | Immediate
  Decrease in amplitude > 25%
Pacing lead threshold | Immediate
  Threshold increase > 0.5 V at a fixed pulse width of 0.4ms
Adverse event | Immediate
  An adverse clinical event

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M Aquilina, MD, Principal Investigator — University Hospital
Locations (1):
- University Hospital, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No